CLINICAL TRIAL: NCT05911932
Title: Investigating Genetic Status in Patients Presenting to Clinic
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Elizabeth Finger, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: 121760
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Dementia, Frontotemporal; Alzheimer Dementia (AD); Lewy Body Dementia (LBD)
Keywords: Neurodegenerative disorders
MeSH Terms: conditions — Frontotemporal Dementia; Alzheimer Disease; Lewy Body Disease; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To examine genetic and polymorphism biomarkers via a blood sample, where the biosample will be tested for genes thought to be relevant to neurodegenerative diseases, and could be re-tested as newly discovered genetic mutations or polymorphisms are revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biosample collection. — Blood draw.

SUMMARY:
The causes of neurodegenerative dementias such as Frontotemporal Dementia, Lewy Body Disease and Alzheimer's disease are still largely unknown. While the contribution of some genetic mutations and polymorphisms is associated with autosomal dominant patterns of inheritance of these dementias, in many cases, the specific causative mutation in these families is not yet identified. Further, in many patients, polygenic risk is thought to give rise to pathophysiologic changes, but which specific genes affect risk are largely yet unknown. By examining genotypes in patients that present to our Cognitive Neurology and Alzheimer's Research Clinic with suspected or confirmed neurodegenerative dementia, or have a history of a familial dementia, we aim to help identify and characterize genetic mutations or polymorphisms that give rise to neurodegenerative diseases.

ELIGIBILITY:
Inclusion Criteria:

* Persons presenting to the cognitive clinic with a neurodegenerative disorder (for example, AD, FTD, LBD, ALSP, and related conditions);
* Biological family members of someone diagnosed with a neurodegenerative disorder, presenting to clinic;
* Age 18+ years old;
* Consenting to a blood draw.

Exclusion Criteria:

• Persons declining / unwilling / not able to have a blood draw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons presenting to the cognitive clinic with a neurodegenerative disorder (for example, AD, FTD, LBD, ALSP, and related conditions);
  Biological family members of someone diagnosed with a neurodegenerative disorder, presenting to clinic;
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2038-08 (Estimated); Study Completion 2043-08 (Estimated)

PRIMARY OUTCOMES:
Blood draw for genetic status or polymorphism result. | A one-time visit, taking the participant approximately 20 minutes total for all study procedures.
  The blood draw is taken at the time of the clinic visit. Up to 30ml will be collected by standard venipuncture.

SECONDARY OUTCOMES:
Demographic information. | A one-time visit, taking the participant approximately 20 minutes total for all study procedures.
  Demographic information will be collected at the time of the clinic visit.
Medical history/Clinical diagnoses. | Typically within 1 month of the clinic visit, taking approximately 5 minutes.
  Will be obtained via chart review when available. This information is collected already as part of the patient's standard care.
Pathological diagnoses. | Typically within 1 month of the clinic visit, taking approximately 5 minutes.
  Will be obtained via chart review when available. This information is collected already as part of the patient's standard care.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Finger, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Parkwood Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No